CLINICAL TRIAL: NCT03345693
Title: Analysis of the Use of Assistive At--Home Hand- Tracking Technology, MoTrack Therapy, in Hand Rehabilitation
Brief Title: Use of MoTrack Therapy in At-Home Hand Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB00106559
Record Dates: First submitted 2017-11-08; First posted 2017-11-17 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2020-07

CONDITIONS: Hand Injuries
Keywords: Rehabilitation; MoTrack Therapy; Telemedicine; Computer Vision; Compliance
MeSH Terms: conditions — Hand Injuries; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treated with MoTrack Therapy (Experimental): Patients receive the MoTrack Therapy device to assist them in their at-home therapy exercises. The patient is instructed to use the MoTrack Therapy device when they want to do their at-home therapy exercises. The patients therapy in the clinic is not affected.
  Interventions: Device: MoTrack Therapy

INTERVENTIONS:
Device: MoTrack Therapy — A software that runs on a tablet or computer that reads information from a Universal Serial Bus external sensor and instructs patients in their exercises, giving patients feedback as necessary, and recording patient progress and activity.

SUMMARY:
This study focuses on the use of a specific type of at-home hand rehabilitation software, MoTrack Therapy, in improving the treatment of hand and wrist injuries.

DETAILED DESCRIPTION:
Compliance of patients to their prescribed at-home exercises is a large issue. To many patients, the exercises are seen as mundane and boring, decreasing the motivation of patients to complete their exercises. However, even when patients do complete their exercises, patients may have difficulty knowing whether the participants are doing their at-home exercises correctly and to the right amount. After leaving his or her therapist's office, the patient usually has nothing more than a written handout, if anything, to guide them through their at-home exercises. Especially since range of motion and pain levels can change daily, it is difficult to expect the patient to consistently do his or her exercises every time, much less to do them correctly. Ineffective exercises and / or a lack of compliance can lead to setbacks, complications, or even expensive and painful repeat surgeries. And at the therapist's office, the therapist may have trouble telling whether setbacks or lack of progress is because of lack of compliance, ineffective exercises, or an underlying medical problem.

Advances in technology have made it possible to track the hands of patients suffering from hand and wrist medical conditions as patients do their at-home exercises. Furthermore, this data can be analyzed in real-time to determine if and how the patient is doing his or her exercises. Another advantage of tracking the hand is that the therapy exercises can be incorporated into a fun computer game that motivates the patient to actually complete their therapy. The hypothesis is that having a computer and accompanying sensors track the hand to give real-time feedback, monitor improvements over time, and gamify the therapy experience to motivate the patient will improve the standard of care given to patients. If this hypothesis is true, patients will understand their exercises better, be inclined to do them more often, and thus have better outcomes. Not only will patients benefit, but the therapist's job will be easier as well. The therapist will have quantitative data to help distinguish medical issues from exercise issues. Ideally, a very successful trial would even suggest a possibility for the patient to rely less on the therapist for the at-home exercises, giving the therapist time to focus on more difficult cases. This research therefore is important because the problems with at-home therapy may be mitigated or solved with such an aid.

ELIGIBILITY:
INCLUSION CRITERIA

* Participants with hand and wrist conditions that require at-home exercises of wrist/finger movements, including dorsiflexion, palmar flexion, radial deviation, ulnar deviation, supination, pronation, thumb adduction, etc.
* Participants who have fractures and similar conditions as the cause of the problem
* Participants must be able to give their own consent.

EXCLUSION CRITERIA

* Pregnant women
* Participants not fluent in English
* Participants below the age of 18
* Participants institutionalized or incarcerated
* Participants who's hand condition is primarily nerve-related as opposed to being caused by a fracture or similar condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Compliance | At the conclusion of the patient's physical therapy (approximately 3 months after starting use of device)
  The software is able to record when the patient is using it, and thus will know how often patients are completing their exercises. The degree to which patients follow their therapist's recommended exercise schedule will be measured.

SECONDARY OUTCOMES:
Patient Ability to Understand the Prescribed Exercises From the Device | Approximately two weeks after patient starts to use the device
  At therapy appointments during the study, patients will be asked to do the exercises with no visual or instructional aid in order to determine if they have learned to do the exercises correctly. If necessary, the patient will be given the software as an aid in order to determine if the patient is then able to complete the exercises.
Prediction of Patient Improvement | Approximately two weeks after patient starts to use the device
  Physical therapy should increase the patient's medical condition over time. In this outcome measure, the ability of the software to predict the patient's improvements in medical condition will be determined by comparing the software predictions of improvement with the actual patient improvements as determined by physical therapists. Medical condition in this case will be operationalized as the extent to which a patient can complete standard hand therapy exercises as measured by the therapist using goniometry.
Prediction of Patient Improvement | Approximately four weeks after patient starts to use the device
  Physical therapy should increase the patient's medical condition over time. In this outcome measure, the ability of the software to predict the patient's improvements in medical condition will be determined by comparing the software predictions of improvement with the actual patient improvements as determined by physical therapists. Medical condition in this case will be operationalized as the extent to which a patient can complete standard hand therapy exercises as measured by the therapist using goniometry.
Prediction of Patient Improvement | Approximately six weeks after patient starts to use the device
  Physical therapy should increase the patient's medical condition over time. In this outcome measure, the ability of the software to predict the patient's improvements in medical condition will be determined by comparing the software predictions of improvement with the actual patient improvements as determined by physical therapists. Medical condition in this case will be operationalized as the extent to which a patient can complete standard hand therapy exercises as measured by the therapist using goniometry.
Prediction of Patient Improvement | At the conclusion of the patient's physical therapy (approximately 3 months after the patient starts using the device)
  Physical therapy should increase the patient's medical condition over time. In this outcome measure, the ability of the software to predict the patient's improvements in medical condition will be determined by comparing the software predictions of improvement with the actual patient improvements as determined by physical therapists. Medical condition in this case will be operationalized as the extent to which a patient can complete standard hand therapy exercises as measured by the therapist using goniometry.
Patient Hand Recovery | Baseline (defined as the therapist visit before the patient starts to use the device) and at the conclusion of the patient's physical therapy, approximately 3 months.
  Using the bMHQ (Brief Michigan Hand Questionnaire), the patient's current state of the hand will be measured. The bMHQ is scored from 0-100, with higher scores indicating better functioning and satisfaction with the hand.The change in the survey results between the first baseline and subsequent measurement represents patient recovery.
Patient Hand Recovery | Baseline (defined as the therapist visit before the patient starts to use the device) and at the halfway point in the patient's expected physical therapy, which is approximately 6 weeks after baseline
  Using the bMHQ (Brief Michigan Hand Questionnaire), the patient's current state of the hand will be measured. The bMHQ is scored from 0-100, with higher scores indicating better functioning and satisfaction with the hand.The change in the survey results between the first baseline and subsequent measurement represents patient recovery.
Patient Satisfaction | At the end of the patient's physical therapy (approximately 3 months after starting use of device)
  The patient will be asked "To what degree did you enjoy doing the exercises, and what feedback do you have for improving the app?". The patient's verbal responses will be recorded. The patient can also express their satisfaction to the investigators anytime during the study as they find criticism.
Therapist Satisfaction | At the end of the patient's physical therapy (approximately 3 months after starting use of device)
  The therapist will be asked "To what degree do you believe the MoTrack device is easy to use with your patients, and what feedback do you have for improving the app?". The therapist's verbal responses will be recorded. The therapist can also express their satisfaction to the investigators anytime during the study as they find criticism.

CONTACTS AND LOCATIONS:
Overall Officials: Scott S Lifchez, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No